CLINICAL TRIAL: NCT00126269
Title: A Randomized Phase III Trial Comparing Cisplatin With or Without Gemcitabine in Patients With Carcinoma of Unknown Primary and a Predicted Favorable Prognosis
Brief Title: Trial Comparing Cisplatin With or Without Gemcitabine in Patients With Carcinoma of Unknown Primary
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEFCAPI O2
Record Dates: First submitted 2005-08-02; First posted 2005-08-03 (Estimated); Last update posted 2006-09-08 (Estimated); Status verified 2006-09

CONDITIONS: Carcinoma
Keywords: Patients with Carcinoma of Unknown Primary and a Predicted Favorable Prognosis
MeSH Terms: conditions — Carcinoma | interventions — Cisplatin; Gemcitabine

INTERVENTIONS:
Drug: cisplatin
Drug: gemcitabine

SUMMARY:
This is a randomized phase III trial comparing cisplatin with or without gemcitabine in patients with carcinoma of unknown primary and a predicted favorable prognosis.

The purpose of this trial is to compare the overall survival rates of patients with carcinoma of unknown primary (CUP) and a predicted favorable prognosis according to the French classification treated with cisplatin with or without gemcitabine.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Evidence of CUP based on histologic examination
* Negative search for the primary tumor site using recommended guidelines
* Disease classified as good prognosis according to the French classification criteria: *performance status >2 and *normal serum LDH
* No prior chemotherapy
* No previous carcinoma, except basal-cell carcinoma of the skin
* Adequate renal function: measured or calculated creatinine clearance > 60 ml/min
* Absolute granulocyte count ≥ 1,500/mm3; platelets ≥ 100,000 mm3; bilirubin ≤ 1.5 fold the upper normal value
* Signed informed consent

Exclusion Criteria:

* Patients infected by the Human Immunodeficiency Virus (HIV)
* CUP belonging to one of the following subgroups: 1) Axillary lymph node of an adenocarcinoma in a woman; 2) Serous adenocarcinoma of the peritoneum in a woman; 3) Undifferentiated carcinoma of the middle line in a young man; 4)Squamous-cell carcinoma; 5) Neuroendocrine carcinoma; 6) Bone metastases with elevated serum prostate specific antigen (PSA) in a man
* Patients who do not fit inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192
Dates: Start 2003-05

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Response rate
Progression-free survival
Toxicity
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Karim FIZAZI, Dr, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, France